CLINICAL TRIAL: NCT03344497
Title: Animated Video Consultation for Reducing Pre-Operative Anxiety in Outpatient Dermatologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1702192435
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2017-11

CONDITIONS: Dermatology/Skin - Other

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VC (Conventional Consultation/Video) Group (Other): Subjects will receive conventional consultation and watch an animated video.
  Interventions: Other: VC Group
- CC (Conventional Consultation) Group (No Intervention): Subjects will receive conventional consultation only. Subjects will cross-over to receive animated video at the end.

INTERVENTIONS:
Other: VC Group — VC (Conventional Consultation/Video) Group
  Arms: VC (Conventional Consultation/Video) Group

SUMMARY:
The purpose of this study is to evaluate whether the addition of an animated skin surgery educational video to conventional in-person surgery consultation will help reduce pre-operative anxiety in patients awaiting outpatient skin surgery.

DETAILED DESCRIPTION:
This will be an randomized controlled pilot study. Subjects will be randomized to either receive an animated video along with conventional consultation OR receive a conventional consultation only. Pre-operative anxiety will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female, at least 18 years of age
2. Subjects scheduled to undergo outpatient skin surgery
3. Subjects able to comprehend and read the English language.

Exclusion Criteria:

1. Subjects unable to or unwilling to comply with the study procedures
2. Subjects unable to speak or read the English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Pre-operative anxiety levels assessed via questionnaire | 1 day
  Preoperative anxiety and information scale will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona - Banner University Medicine Dermatology, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No